CLINICAL TRIAL: NCT05376488
Title: Characterization of Venous Ammonia Levels in Fasted and Fed State in Patients With Cirrhosis After Vegetarian, Vegan and Non-Vegetarian Meals
Brief Title: Effect of Brief Dietary Intervention on Ammonia Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: BAJAJ030
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Cirrhosis; Hepatic Encephalopathy
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy

STUDY DESIGN:
Intervention Model Description: Randomized single blind
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meal type A (Active Comparator): Meal type A: equicaloric meal as meal type B and C with differing constituents
  Interventions: Other: One meal
- Meal type B (Active Comparator): Meal type B: equicaloric meal as meal type A and C with differing constituents
  Interventions: Other: One meal
- Meal type C (Experimental): Meal type C: equicaloric meal as meal type B and A with differing constituents
  Interventions: Other: One meal

INTERVENTIONS:
Other: One meal — One meal given to assess impact on ammonia levels serially

SUMMARY:
Study the impact of differing meal contents on venous ammonia levels over time in patients with cirrhosis. Patients will be given specific meals and venous ammonia analyzed over time after those meals.

The subjects will also provide stool for microbiome and serum, urine and plasma for metabolomics during this one-time study.

Total duration=4 hours

DETAILED DESCRIPTION:
Patient will be instructed to collect stool for baseline assessments. After a fast (>4h from last meal) a venous blood sample will be drawn for analysis of baseline laboratory tests and spot venous ammonia and blood and urine for metabolomics and blood microbiome. Spot ammonia and blood for metabolomics and microbiome will be collected from repeat samples at 1h and 2 hrs after a standardized meals from the three groups of protein meals. Urine will also be collected for metabolomics during the observation period. On the day of the study, patients will be asked to complete a standard food frequency questionnaire encompassing meals over 3 days prior to the study.

Subjects will be randomly assigned into 3 groups (meal types A, B and C) with the standardized meal that contains 20gm of protein. All subjects are expected to consume it in its entirety. Subjects are not allowed to eat anything else until the end of the study.

Subjects will be observed in the unit for a total of 3 hours after the standardized meal to ensure no symptoms related to potential elevated ammonia emerge. Any adverse events will be treated according to standard clinical routine.

ELIGIBILITY:
Inclusion Criteria:

1. Cirrhosis
2. Able and willing to voluntarily complete the informed consent process
3. Available for and agree to all study procedures
4. Consistent non-vegetarian Western dietary patterns for at least a month prior to the study assessed by dietary interview

Exclusion Criteria:

1. MELD score > 23
2. Unclear diagnosis of cirrhosis
3. History of liver transplant
4. Body mass index < 18.5 or ≥ 40 kg/m2
5. Prior transjugular intrahepatic portosystemic shunt placement
6. Treatment with systemic (e.g., oral or intravenous) antibiotic (apart from rifaximin) within 4 weeks prior to enrollment
7. For those with HE: stable dose of medications (lactulose or rifaximin) without a recent (<1 month episode of HE)
8. Current use of valproate, corticosteroids, or cytotoxic drugs.
9. Apart from chronic liver disease, any acute or chronic medical, surgical, psychiatric, or social condition including history of cerebrovascular disease (stroke, transient ischemic attack) or dementia, that may increase the subject risk associated with study participation, compromise adherence to study procedures and requirements, confound interpretation of the results, and, in the judgment of the investigator, make the subject inappropriate for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Venous ammonia level | 3 hours
  Change in these levels hourly from baseline

SECONDARY OUTCOMES:
Venous ammonia level | 1 hour
  Change in these levels from baseline to hour 1
Venous ammonia level | 2 hours
  Change in these levels from baseline to hour 2
Venous ammonia level | 3 hours
  Change in these levels from baseline to hour 3

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan Bajaj, Principal Investigator — Hunter Holmes McGuire VAMC
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT05376488/ICF_000.pdf